CLINICAL TRIAL: NCT05769686
Title: LAParoscopic DOnor nephreCTomy scORe (LAPDOCTOR) Multicenter Validation of a New Scoring System for Preoperative Prediction of Difficulty of Laparoscopic Donor Nephrectomy
Brief Title: Laparoscopic Donor Nephrectomy Score, a New Scoring System for Preoperative Prediction of Difficulty of Laparoscopic Donor Nephrectomy
Acronym: LAPDOCTOR
Status: Completed | Type: Observational
Sponsor: Jacopo Romagnoli (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Ospedaliera di Padova (Other); Ospedale Pediatrico Bambin Gesù (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Ospedaliera Niguarda Cà Granda (Other)
Responsible Party: Sponsor-Investigator, Jacopo Romagnoli, Surgical Director Renal Transplant Unit, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Organization: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Other Study IDs: 2939
Record Dates: First submitted 2023-02-16; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Renal Failure Chronic; Surgery
Keywords: living donation; laparoscopic nephrectomy; difficulty; scoring system
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this multicenter observational study is to develope and validate a new scoring system for preoperative prediction of difficulty of Laparoscopic Donor Nephrectomy. Healthy living kidney donors will be enrolled. The main questions it aims to answer are: 1) can the investigators predict difficulty of the operation ? 2) Can the investigators score difficulty based on this new scoring system? Difficulty of LDN will be graded by the operating surgeon at the end of the operation based on intraoperative predefined parameters. All operations will be blindly scored by the operating surgeon, while one radiologist will blindly review all preoperative CT scans. LAPDOCTOR scores will be compared with the degrees of difficulty assigned by the operating surgeon to investigate the match rate.

DETAILED DESCRIPTION:
The LAPDOCTOR scoring programme calculates the score based on presence, absence of certain characteristics (Sex, BMI, different radiologic measurements, etc.). A score of 1 to 2 is assigned to each characteristics . Difficulty is graded as standard when the sum is between 11 and 18, moderately difficult between 19 and 25, very difficult between 26 and 33). At the end of the operation the donor surgeon will score the difficulty assigning a score of 1 to 3 to each phase of the operation, the resulting score will define again three degree of difficulty (standard 1-8, moderately difficult 9-16, very difficult 17-24.

ELIGIBILITY:
Inclusion Criteria:

- Age of donor ≥ 18 yrs (minimum 18, maximum , deemed suitable for donation at the end of work-up

Exclusion Criteria:

* age< 18 yrs
* hypertension with organ damage
* unable to express proper consent to procedure
* evidence of coercion
* drug abuse
* evidence of malignancy
* pregnancy
* major respiratory or cardiovascular risk
* diabetes mellitus
* renal disease
* systemic disease with renal involvement
* thrombophilia
* BMI >35
* active infection
* hepatitis B, hepatitis C and HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Candidates to living kidney donation
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of donors with a score between 26 and 33 in the LADOCTOR scale (risk of very difficult operation) | 12 months
  The LAPDCOTOR scoring programme calculates the score based on presence, absence of certain characteristics (Sex, BMI, different radiologic measurements, etc.). A score of 1 or 2 is assigned to each characteristics . Difficulty is graded as standard when the sum is between 11 and 18, moderately difficult between 19 and 25, very difficult between 26 and 33).

SECONDARY OUTCOMES:
change in intraoperative complications | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacopo Romagnoli, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Policlinico Universitario A. Gemelli, Rome, Lazio, Italy

REFERENCES:
- [Derived] Romagnoli J, Spagnoletti G, Rossini FE, Iezzi R, Posa A, Salerno MP, Silvestri P, Rossini AE, Silvestre C, Franchin B, Giacomoni A, Centonze L, Spada M, Iaria M, Puliatti C, Furian L. Lapdoctor: Multicentre Validation of a Scoring System for Preoperative Evaluation of Difficulty of Laparoscopic Donor Nephrectomy. Transpl Int. 2025 Apr 23;38:14100. doi: 10.3389/ti.2025.14100. eCollection 2025. PMID 40336540